CLINICAL TRIAL: NCT04534998
Title: ROBOtic-assisted Versus Conventional Open Partial Nephrectomy: a Single-center, Open-label, Randomized Controlled Feasibility Trial
Brief Title: Robotic-assisted vs. Open Partial Nephrectomy
Acronym: ROBOCOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Institute of Medical Biometry and Informatics, University of Heidelberg (Unknown); Dietmar Hopp Stiftung (Other)
Responsible Party: Principal Investigator, Karl-Friedrich Kowalewski, Principal Investigator, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-542N
Record Dates: First submitted 2020-08-16; First posted 2020-09-01 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic-assisted partial nephrectomy (Experimental): Partial nephrectomy will be performed using a robotic-assisted laparoscopic approach.
  Interventions: Procedure: Partial nephrectomy
- Open partial nephrectomy (Active Comparator): Partial nephrectomy will be performed using an open retroperitoneal approach.
  Interventions: Procedure: Partial nephrectomy

INTERVENTIONS:
Procedure: Partial nephrectomy — Partial nephrectomy for localized kidney cancer as curative treatment.
  Other Names: nephron-sparing surgery

SUMMARY:
ROBOCOP is an open-label, randomized controlled feasibility trial comparing robotic-assisted and open partial nephrectomy in preparation for a confirmative phase III randomized controlled trial.

DETAILED DESCRIPTION:
Surgical excision is the gold standard for the treatment for localized kidney cancer. An organ-preserving procedure should be carried out whenever possible in order to maintain kidney function. Partial nephrectomy can be performed through the conventional open technique as well as through a robotic-assisted approach. Although both methods belong to the standard care, there is still no published data from randomized controlled trials in the scientific literature comparing them. The ROBOCOP-trial is designed as a single-center comparison of the two surgical approaches in preparation for a phase III study. 50 patients are to be included in the trial within a period of 15 months. The primary endpoint is feasibility of patient recruitment. In addition, potential primary outcomes for a confirmative trial such as perioperative complications, quality of life, inflammatory response, survival and ergonomic aspects for the operating surgeons will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective partial nephrectomy for renal neoplasms
* Patient must be at least 18 years old and capable to consent
* abdominal MRI or CT scan
* curative-intent surgery
* robotic-assisted and open approach for surgery are both feasible
* ability of patient to understand the goal, consequences and alternatives of participation in the trial
* written informed consent

Exclusion Criteria:

* patients with solitary kidney
* multiple kidney tumors
* emergency intervention, for example because of bleeding or perforation
* 2nd malignancy that will make PN needless, this does not include secondary malignancies which are under curative treatment or cases in which death from RCC is more likely
* patient belongs to a vulnerable patient group
* simultaneous 2nd surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 15 months
  Proportion of randomized patients in relation to the eligible ones.

SECONDARY OUTCOMES:
Perioperative complications | throughout patient´s hospital stay, on average 6 days
  Measured with 1) the comprehensive complication index (CCI), on a scale from 0 (no complications) to 100 (death) and 2) the Clavien-Dindo classification, which consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V), the first one indicating any deviation from the normal postoperative course, the highest grade indicating death
Postoperative complications | 90 days
  Measured with 1) the comprehensive complication index (CCI), on a scale from 0 (no complications) to 100 (death) and 2) the Clavien-Dindo classification, which consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V), the first one indicating any deviation from the normal postoperative course, the highest grade indicating death
Self-reported generic health status | 90 days
  Patient-reported generic health status using EQ-5D-5L(EuroQol-5D-5L) questionnaire (the scale ranges from 0 to 100, with 100 representing the highest health status)
Self-reported quality of life assessment of cancer patients | 90 days
  Cancer patients will be reporting their quality of life making use of the questionnaire QLQ-C30 (Quality of Life Questionnaire C30) (range 0-100, high scores represent a better quality of life)
Self-reported quality of life in patients with kidney disease | 90 days
  Patients will assess the influence of their kidney disease on everyday activities, work status, social interactions, mental and physical health making use of KDQOL-SF (Kidney Disease Quality of Life Short Form), ranging from 0 ("worst possible health") to 10 ("best possible health")
Self-assessment of depression in patients ≥ 65 years old | 90 days
  Elderly patients (≥ 65 years old) will report their depression symptoms filling GDS (Geriatric Depression Scale) questionnaire, ranging from 0 to 30, with 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Self-evaluation of cancer disease´s influence on elderly patients´ life | 90 days
  Elderly patients (≥ 65 years old) will evaluate the influence of their cancer disease on their life (activities of daily living, cognition, mood, nutritional status, mobility, polypharmacy and social support), on a scale ranging from 0 to 17, 17 indicating the best outcome possible on quality of life.
Self-assessment of comorbidity in elderly patients | 90 days
  Elderly patients (≥ 65 years old) will make use of SCQ (Self-Administered Comorbidity Questionnaire) to assess common comorbidities; a higher score indicates higher comorbidities (range 0-39)
Postoperative self-reported quality of life | 90 days
  Participants will evaluate their postoperative quality of life on a 0-100 scale, higher scores indicating a better quality of life and return to daily life activities.
Kidney function - creatinine | 90 days
  postoperative change in kidney function - creatinine (measured in mg/dL)
Kidney function - GFR | 90 days
  postoperative change in kidney function - glomerular filtration rate (measured in mL/min)
Length of hospital stay | throughout patient´s hospital stay, on average 6 days
  Total time of hospital stay
Operative time | Immediately after surgery
  Surgery duration
Inflammatory response - leucocytes | throughout patient´s hospital stay, on average 6 days
  postoperative course of inflammatory parameters (leucocytes, unit of measure: white cells x10^9/L)
Inflammatory response - C-reactive protein | throughout patient´s hospital stay, on average 6 days
  postoperative course of inflammatory parameters (c-reactive protein, measured in mg/L)
Inflammatory response | throughout patient´s hospital stay, on average 6 days
  postoperative course of inflammatory parameters (IL-6, TNF-α, IL-1β, VEGF, measured in ng/L)
Surgical ergonomics | Immediately after surgery
  Surgeons will be asked to evaluate localized muscle pain on a scale from 0 to 10, 10 indicating extreme discomfort
Surgical ergonomics | During surgery
  Surgeons will be asked to fill NASA TLX questionnaire (NASA Task Load Index). Range: 0-100, high scores indicate a high task load
Resection status | up to 5 days
  Rate of R0/R1 status in each arm
Use of analgesia | throughout patient´s hospital stay, on average 6 days
  Need for pain medications
Trifecta outcomes of partial nephrectomy | 90 days
  Trifecta is defined as no major complication, R0-resection status and ischemia time of less than 25 minutes
Blood loss | Immediately after surgery
  Blood loss during surgery
Conversion to open surgery | Immediately after surgery
  Rate of conversion to open surgery
Conversion to radical nephrectomy | Immediately after surgery
  Rate of conversion to radical nephrectomy
Case cost | 90 days
  DRG-related case costs per arm

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian C. Kriegmair, M.D., Study Director — Department of Urology, University Medical Center Mannheim, University of Heidelberg
Locations (1):
- Department of Urology, University Medical Center Mannheim, University of Heidelberg, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient information might be shared after signing a data sharing agreement and IRB approval
Supporting Information: Study Protocol, Analytic Code
Time Frame: After completion of the study (anticipated March 2021)

REFERENCES:
- [Derived] Kowalewski KF, Sidoti Abate MA, Neuberger M, Kirchner M, Krisam R, Egen L, Haney CM, Siegel F, Michel MS, Honeck P, Nuhn P, Westhoff N, Kriegmair MC. ROBOCOP II (ROBOtic assisted versus conventional open partial nephrectomy) randomised, controlled feasibility trial: clinical trial protocol. BMJ Open. 2021 Nov 3;11(11):e052087. doi: 10.1136/bmjopen-2021-052087. PMID 34732486